# RESEARCH PARTICIPATION INFORMATION AND CONSENT FORM For Protocol Addendum #2

**TITLE:** A virtual Phase 2 randomized, placebo-controlled, double

blind study to evaluate the safety and efficacy of the

combination of famotidine and celecoxib as a post-exposure prophylaxis (PEP) for newly infected COVID-19 patients

**SUB-STUDY TITLE:** A virtual Phase 2 randomized, placebo-controlled, double-

blind study to evaluate the safety and efficacy of the combination of famotidine and celecoxib with and without ivermectin as a post-exposure prophylaxis (PEP) for newly-

infected COVID-19 patients

**SHORT TITLE:** LEAP-CT for evaluation of post-exposure prophylaxis for

newly-infected COVID-19 patients

PROTOCOL NO.: LDOS-21-001-02

IND 153669

WCG IRB Protocol #20211500

**SPONSOR:** Leidos, Inc.

**FUNDING** 

**ORGANIZATION:** United States Department of Defense (DoD)

Defense Threat Reduction Agency (DTRA)

<<CF-Main Header Block - Investigator>>

**INVESTIGATOR:** Name

Address

City, State Zip

Country

STUDY-RELATED

PHONE NUMBER(S): << CF-Main User Defined #1>>

Phone Number

Phone Number (24 hours)
[24-hour number is required]


#### INFORMED CONSENT SUMMARY

You are being asked for your consent to take part in a research study. This document provides a concise summary of this research. It describes the key information that we believe most people need to decide whether to take part in this research. Later sections of this document will provide all relevant details.

#### What should I know about this research?

- Someone will explain this research to you.
- Taking part in this research is voluntary. Whether you take part is up to you.
- If you don't take part, it won't be held against you.
- You can take part now and later drop out, and it won't be held against you.
- If you don't understand, ask questions.
- Ask all the questions you want before you decide.

# How long will I be in this research?

We expect that your taking part in this research will last 90 days.

#### Why is this research being done?

The purpose of this research is to study whether an investigational combination of famotidine (commonly used to treat heartburn) and celecoxib (commonly used to treat arthritis) can improve symptoms in people who are newly diagnosed with COVID-19, showing mild symptoms.

#### What happens to me if I agree to take part in this research?

If you decide to take part in this research study, the general procedures include taking the study drugs or placebos, measuring your heart function with a mobile electrocardiogram (ECG), getting your blood drawn, and answering questionnaires.

#### Could being in this research hurt me?

The most important risks or discomforts that you may expect from taking part in this research include risks from famotidine (headache, dizziness, constipation, diarrhea, kidney injury) and celecoxib (abdominal pain, diarrhea, upset stomach, swelling, dizziness, sore throat, rash, kidney injury, and liver injury).


### Will being in this research benefit me?

The most important benefit that you may expect from taking part in this research include improvement of your symptoms from COVID-19. However, this cannot be promised. Possible benefits to others include learning about another treatment for COVID-19.

# What other choices do I have besides taking part in this research?

Instead of being in this research, your choices may include other medications used to treat COVID-19, like remdesivir, baricitinib and dexamethasone if you are in the hospital; monoclonal antibodies and/or antiviral treatments that have been granted Emergency Use Authorization (EUA) from the US Food and Drug Administration (FDA), for those who qualify; supportive care; and joining another research study.

#### INFORMED CONSENT FORM

You are being asked to participate in an on-line (virtual) clinical research study that seeks to find a possible treatment for COVID-19. Please take your time to read this consent form so that you understand the purpose, risks, and benefits. Taking part in this study is voluntary.

We urge you to ask any questions you might have of the study team, and to make your decision thoughtfully. If you decide to participate, you must sign this form to show that you want to take part.

#### Why is this research study being done?

Coronavirus disease 2019 (COVID-19) is a highly infectious virus (called coronavirus, or SARS-CoV-2) that was newly discovered in 2019. It has spread rapidly around the world causing a global pandemic, and millions of people have become very sick. You are being asked to take part in this study because you have either recently tested positive for COVID-19, or you suspect that you have the illness and are waiting for the results of a laboratory test. You are likely experiencing mild symptoms, but can still perform daily tasks. People who have COVID-19 may have flu-like symptoms such as cough, shortness of breath, nausea, and feeling tired, fever, chills, muscle stiffness, headache, sore throat, and/or loss of smell.

Right now, there are two FDA approved treatment for COVID-19 in hospitalized patients – Remdesivir (Veklury®), Olumiant® (baricitinib). Some monoclonal antibody and/or antiviral therapies have been granted an EUA for the treatment of mild to moderate COVID-19 symptoms may be available to people 12 years of age or older with positive results of direct SARS-CoV-2 viral testing, and who are at high risk for progressing to severe COVID-19, including hospitalization and death.


There is a critical need to find medications that can slow down or stop COVID-19 from damaging the body. The purpose of this research study is to learn more about two (2) FDA-approved drugs that are currently available on the market and used to treat other conditions. The two drugs used in this study are not approved by the FDA to treat COVID-19. They *might* help prevent people with a mild case of COVID-19 from getting sicker, having to be hospitalized, or dying.

We want to test these drugs together to see if the combination helps prevent COVID-19 from getting worse in people with mild cases of the disease. We also want to learn about any unknown side effects that might happen after taking the study medications together, and at doses that are different from what is usually prescribed. Since these drugs have not been used in combination to treat COVID-19 before, they are considered investigational. The two drugs that we want to learn more about are:

| Study Drug Name | Common Name | Current Uses |
|-----------------|-------------|------------------|
| Famotidine | Pepcid AC® | Treats heartburn |
| Celecoxib | Celebrex® | Treats arthritis |

Some people die from COVID-19 because of the body's reaction to the virus. In some cases of COVID-19, people will experience a *hyper*-inflammatory response where the body begins to attack the virus, but overreacts by attacking the healthy parts of the body. Each of the drugs that we are studying show some proof that they reduce inflammation and that they can work by themselves to treat the inflammation in different ways. This study seeks to learn whether these drugs help reduce the hyper-inflammatory response that is triggered by SARS-CoV-2 infection.

You have been asked to participate in this study because you have a confirmed or suspected case of COVID-19 with mild symptoms. We want to see if these two drugs are safe to use together, and we want to see how the study drugs affect your symptoms. We also would like to keep track of your symptoms, using an online questionnaire before and after you take the study drugs. We want to see if the combination of these drugs (famotidine and celecoxib) will diminish your symptoms and/or reduce the time it takes for you to feel better.

### What will happen during the study if I agree to participate?

In this study, you will be assigned, or "randomized," into one of the two (2) study groups described below. "Randomized" means that you are put into a group by chance, like flipping a coin. You will have an equal chance of being placed in either group. It is important to know that this study is "double-blinded," meaning that neither you nor the study doctor or the study staff will know which group you are in until after the study has ended. In the event of an emergency, this information can and will be made available.

| Group | Study Drug Regimen |
|---|---|
| Group 1: You will receive the two (2) study drugs | <ul> <li>80 mg of famotidine taken by mouth 4 times per day for 5 days with</li> <li>A one time, first dose of 400 mg of celecoxib on the first day, then 200 mg of celecoxib taken by mouth 2 times per day for 5 days</li> <li>After the completion of the 5-day treatment course, you will continue taking famotidine 4 times per day for 9 more days.</li> </ul> |
| Group 2: You will receive a placebo of each study drug | <ul> <li>A placebo taken by mouth 4 times per day for 5 days with</li> <li>A placebo taken by mouth 2 times per day for 5 days.</li> <li>A placebo taken by mouth for 9 days</li> </ul> |

Placebo: This means that you will receive medication that looks exactly like the drugs that are being studied but only contains inactive substances that have no treatment effect or therapeutic value.

There will be approximately 1800 people evaluated to take part in this study from across the United States, and about 1450 who join the study after being evaluated. Your participation is voluntary, and you have the alternative to not take part in this research study. You may discuss other treatments for COVID-19 and management of COVID-19-related symptoms and reactions with the study doctor or your treating physician.

If you decide to take part in this study, your participation will include the following:

You will be asked to answer questions on your personal electronic device (e.g., a cell phone, tablet or computer) to see if you can participate in the study. You will also be asked to:

- Read and sign this informed consent form after a virtual discussion with the study doctor(s);
- Provide information about your medical history;
- Provide information about the medications and supplements you take.
- Provide an initial blood sample of 10mL 15mL (about 2-3 teaspoons).
- Provide the results from your positive PCR test or be swabbed for a PCR test if you took an at-home antigen test.


# LEAP-CT for evaluation of post-exposure prophylaxis for newly-infected COVID-19 patients 18 February 2022

IRB Approved Template MUST BE APPROVED FOR SITES BEFORE USE AS MODIFIED Jul 07, 2022

Once the doctor confirms you are eligible to participate you will be enrolled in the study. You will:

- Receive a package containing your assigned study medications. The package will not tell you which drugs you are being given. You will be asked to confirm with the study doctor that you received the package.
- Be asked to take your medicines each day, as directed;
- Provide 2 additional blood samples (on Day 7 and Day 14) of 10 mL 15 mL (about 2-3 teaspoons);
- Be asked about any new symptoms you're experiencing and how bad they are making you feel (daily, for 90 days);
- Take your temperature and measure your oxygen levels every day for 90 days (You will be provided with the equipment to measure these at no cost to you);
- Utilize a heart function monitor to record a mobile ECG on Day 7 and Day 14;
- Follow-up with your doctor for any health concerns or issues;
- Be evaluated by remote interview with the study doctor (2 months after the first day you take the study drugs and again at 3 months after the first day you started taking the study drugs).

This study will be virtual. This means that you will not physically visit the study doctor in person, and the study drugs will be delivered to your home or designated address. In order to collect the necessary blood samples, a phlebotomist will come to your home 3 separate times, and draw your blood (at screening, Day 7, and Day 14). The phlebotomist will be scheduled through the electronic platform. You will be asked to take the study drugs, and report that you did so at the appropriate times in an online form through a study website (with a secure link designed to protect your privacy). You will be able to access the website on your personal electronic device, such as a cell phone, tablet or laptop. You will also visit this website daily to answer questions about your COVID-19 symptoms, and your general health and well-being. The online questionnaire will take about 5 to 10 minutes to complete every day.

You will be provided with three electronic devices that you will use to collect the necessary data about your body temperature, oxygen levels, and heart function during the study. Your doctor will receive your test results through the website and look at the data. Help is available through the website at all times if you have any issues or questions.

Your participation in this study will last approximately 3 months (90 days).

You can decide to stop taking part in the study at any time. If you decide to stop, let your study doctor know as soon as possible. This is so your study doctor can perform an assessment and talk to you about any follow-up care and testing that could be helpful for you.

# What side effects can I expect from taking part in the study?

You may have side effects while taking the study drugs. Some, but not all, of the common side effects are listed below. Both of the FDA-approved study drugs have a good safety profile and are established as safe for human use when used at the FDA-approved dose for their given indications; however, the dose you may be receiving is more than the FDA-approved dose, and these drugs have never been used together to treat COVID-19.

It is possible that you may experience one or more of the known side effects, or you may experience a side effect that is unknown, or you may experience no side effects at all. Many of these side effects resolve when you stop taking the drugs, but in some cases, the side effects may be serious and/or lasting. Other side effects may be rare, but very serious, and even result in death. The study doctors will not know who will or will not have side effects. You, as the participant, are the only person allowed to take the study drugs as directed. You must keep the study drugs out of the reach of children and persons who might not be able to read or understand that they should not take the study drugs.

#### Famotidine Side Effects:

- Less likely: Fever, nausea, dry mouth, fatigue (or tiredness), dizziness, diarrhea, and/or constipation.
- Rare: Fast/slow/irregular heartbeat, fainting, seizures, rash, bruising/bleeding, and mental/mood changes.

#### Celecoxib Side Effects:

- Less likely: Sore throat, dizziness, gas, diarrhea, and abdominal pain.
- Rare: Rash, severe headache, pain or swelling in the groin or calf, difficulty swallowing, upper respiratory tract infection, kidney injury, liver injury, and serious cardiovascular thrombotic events like myocardial infarction and stroke.

Page **7** of **15** 

#### Celecoxib + Famotidine Side Effects:

There may be unknown side effects from the combination of these two drugs.

### Other Possible Risks Associated with Participating in this Study

**Blood draw risks**: We will be collecting many blood samples from you for evaluation. The risks of drawing blood (venipuncture) include temporary discomfort from the needle stick, bruising, bleeding, and rarely, infection. Blood drawn by trained professionals will help minimize this risk.

**ECG risks:** You will use a mobile device to obtain an ECG at 3 time points during the study and there is very little risk using this FDA-approved device.

**Reproductive risks**: There may be other unknown risks or side effects or discomforts that we cannot predict, especially to an unborn child. Because the drugs in this study may affect an unborn baby, you should not become pregnant or father a baby while on this study. You must use acceptable methods of birth control such as oral contraceptives (the pill), an intrauterine device (IUD), and/or condoms. Your doctor will discuss this with you. You also should not breastfeed a baby while on this study.

**Risk of randomization**: You will be assigned to a treatment group by chance. There is a risk that the treatment you are assigned to may not work as well, or may have more side effects, than the other group. Your condition and/or symptoms may not improve, or may worsen while participating in this study.

**Risks of drug interactions**: The study drug(s) could interact with the other study drugs. These drug interactions could lead to increased side effects. Your study doctor will review all of the drugs and supplements you are currently taking before you start this investigational treatment.

There are some drugs that you cannot keep taking while on the study, and the study doctor will talk to you about. In some cases, you cannot participate in the study if you decide to stay on certain medications.

Risk of collecting a sample of mucus from your nose for a PCR test (a sample will only be collected if you tested positive using an at-home test): The swab used to collect a sample of mucus from your nose is a long flexible stick with a soft tip. You may experience some discomfort including coughing, mild bleeding, or watery eyes.

### What are the benefits of this study if I decide to participate?

You might not receive any direct benefit by participating in this study. If you are randomized into the group that gets the investigational combination of FDA-approved study drugs, there is a chance that your condition and symptoms will improve, but there is no guarantee. The combination of the study drugs was selected because researchers hope that these drugs will help reduce how badly you feel. You will be providing valuable information that may help others who become sick with COVID-19 in the future. We hope the valuable information learned from this study will directly benefit other people by providing a safe and effective treatment for those infected with COVID-19.

A Data Safety and Monitoring Board (DSMB), an independent group of experts, will be reviewing data from this research throughout the study. One of the most important answers we seek to obtain is whether this combination of drugs is not only safe to give, but also whether the doses of the drugs are effective to treat COVID-19. Because we are evaluating the safety and effectiveness of this drug combination, the DSMB will review the data at certain time points, and can be called to meet in case of an emergency. We will tell you in a timely matter about any new information given to us from the DSMB that may affect your health, welfare, or willingness to stay in this study.

# If I choose to participate in the study, can I change my mind later?

Your participation is voluntary, so you can decline to take party in this study. You also may withdraw from the study at any time. Your decisions will not result in penalty or loss of benefits to which you are otherwise entitled. If you decide to withdraw your permission to participate:

- We will no longer use or share medical information about you, or your samples and data, for this research study, except where the law allows us to do so;
- We are unable to delete any information we have already shared with your permission;
- We may continue using and sharing information that was gathered before your withdrawal if it is necessary for the soundness of the overall research;
- We will keep our records of the care we provided to you for as long as required by law.

Your decision not to participate, or to withdraw, will not affect your medical care. Your study doctor will continue to answer any questions you may have, and you will also be advised to see your primary care provider. Alternatively, the study doctor may decide to take you out of the study if new information about the study medication becomes

available that would jeopardize your health and well-being, or if he/she feels it is in your best interest. The study doctor also has the ability to remove you from the study without your consent.

# Will it cost me to participate?

All clinical and professional fees that are associated with this study will be provided at no cost to you. The study medications will also be provided and shipped to your home at no cost. The mobile ECG device, thermometer, and pulse oximeter that are provided will be at no cost to you, and they are yours to keep.

## Will I be paid to participate?

<CF-Main Payment for Part. Paragraph>>For your time, you will be given \$50.00 for each completed study visit, up to a maximum of \$300.00, at the end of the trial (Study Day 90). The study visit payments are as follows:

| Study Visit Number | Study Day | Payment |
|----------------------|---------------------------|------------|
| Screening, Visit 1 | Day -7 to Day -1 | \$50 |
| | Includes a blood draw | |
| Study Visit 2 | Day 1 Baseline/Start of | No payment |
| | Treatment | |
| Study Visit 3 | Day 7 (±1 day) | \$50 |
| | Includes a blood draw | |
| Study Visit 4 | Day 14 (±1 day) | \$50 |
| | Includes a blood draw | |
| Study Visit 5 | Day 30 (±1 day) End of | \$50 |
| _ | Treatment | |
| Study Visit 6 | Day 60 Observation period | \$50 |
| Study Visit 7 | Day 90 Observation period | \$50 |
| (Conclusion of study | - | |
| participation) | | |

When you have completed all study visits, a payment will be made to you in the form of a gift card to the e-mail address you used to register for this study. The total compensation for this study, if you complete all study visits, is up to \$300. If you withdraw or terminate from the study before the end of the study, you will be paid for each visit you completed.

# LEAP-CT for evaluation of post-exposure prophylaxis for newly-infected COVID-19 patients 18 February 2022

IRB Approved Template MUST BE APPROVED FOR SITES BEFORE USE AS MODIFIED Jul 07, 2022

You and/or your insurance plan will need to pay for the standard costs of medical care for treating your condition if needed while participating in the study, just as you would if you were seeking medical care for COVID-19 from your primary care provider.

## What happens if I am injured in this study?

This study is funded by the U.S. Department of Defense (DoD), with Leidos, Inc. acting as the Sponsor for the study on behalf of the DoD. The funder and clinical sites have no plans to pay for any research-related injury, or associated costs that are not covered as part of the study plan. If you are injured in this study, treatment will be provided. If you suffer a study-related injury while participating, Leidos, Inc. will provide reimbursement for the costs of medical treatment.

<<CF-Main Financial Disclosure>>

#### Will my personal information be kept private?

Information gathered in this research study may be published or presented in public forums, but your name and other identifying information will not be used or revealed. Medical records that contain your identity will be treated as confidential. All records will be kept in a locked and secure area and only those persons assigned to this study will have access to those records. All study documents related to you and your participation will show only your assigned patient number (or code). If any of your research records need to be copied, your name and all identifying information will be removed.

Your personal information may also be disclosed if required by law. Despite these efforts to keep your personal information confidential, we cannot guarantee absolute confidentiality. However, your privacy is very important to us, so every reasonable effort will be made to keep your personal information in your research record private and confidential.

Other regulatory groups may become aware of your participation in this study and may require access to your study records in the event of an audit. These groups may include:

- The FDA and the groups it works with to review studies;
- Government agencies, such as the Human Research Protection Office (HRPO) for the US Army Medical Research and Development Command (USAMRDC), involved in keeping research safe for people;
- WCG Institutional Review Board -, a group of people who review the research with the goal of protecting people who take part in the study; <<CF-Main SMO Company 1>><<CF-Main Affiliated IN Language 1>>

- The funders, the DoD & The Defense Threat Reduction Agency (DTRA), and Leidos, Inc., the sponsor of this clinical study;
- Monitoring entities contracted to the sponsor to ensure the trial is done in accordance with FDA regulations, and the data provided from this trial are accurate, and valid.

#### The Use of Private Health Information

Health information about you will be collected if you choose to be part of this research study. Health information is protected by law, as explained in the <<CF-Main User Defined #2>>[Site] Privacy Notice. If you have not received this notice, please request a copy from the study staff. At <<CF-Main User Defined #2>>[Site] your information will only be used or shared as explained and authorized in this consent form, or when required by law. It is possible that some of the other people or groups who receive your health information may not be required by Federal privacy laws to protect your information and may share it without your permission.

To participate in this research you must allow the study team to use your protected health information (PHI). PHI is any information in the medical record or patient file that can be used to identify you, like your name, age, ethnicity, home address, and health status. Federal regulations allow researchers to access and use PHI when necessary to conduct clinical studies. If you do not want us to use your PHI, you may not participate in this study. The research-related therapy is investigational; therefore, it is not available to you unless you allow the use of your PHI.

People usually have a right to access their medical records. However, this research study is blinded. This means that you will not know which treatment group you are in. until after the study has ended. You may receive the drug combination, or you may receive placebo. While this research study is in progress, you may not be allowed to see or copy certain information that is related to this research study. This is only for the period of the research. You will be allowed to see that information when the entire research project is complete.

#### If I have questions or concerns during the study, who do I contact?

You have the right to ask any questions you may have about this research. If you have questions, complaints, concerns, or believe you have developed an injury related to this research, contact <<CF-Main User Defined #3>>[Name] at [Number(s)], or the study doctor on 24 hour call at <<CF-Main User Defined #4>>[Number]. The study doctor will notify the sponsor. You are not waiving any of your legal rights by signing this consent form, nor releasing the sponsor from their legal and professional responsibilities. We will make every effort to prevent injuries or illness from occurring while you are in the study.


If you have questions regarding your rights as a research participant, or you have general questions, complaints or concerns about the research or your privacy and the use of your PHI, contact the research subjects' protection advocate in the <<CF-Main User Defined #2>>[Site] Subjects Protection Office at<<CF-Main User Defined #4>>[Number]. You may also call this number if you cannot reach the research team or wish to talk to someone else.

This research is being overseen by WCG Institutional Review Board (IRB). An IRB is a group of people who perform an independent review of research studies. You may talk to them at or via email at if:

- You have questions, concerns, or complaints that are not being answered by the research team.
- You are not getting answers from the research team.
- You cannot reach the research team.
- You want to talk to someone about the research.
- You have questions about your rights as a research subject.

For more information about participation in a research study, and about the IRB, a group of people who review the research to protect your rights, please visit the WCG IRB's web site at (www.wcgirb.com). Included on this web site, under the heading "Participant Information", you can access Federal regulations and information about the protection of human research participants. If you do not have immediate access to the internet, copies of these Federal regulations are available by calling the <<CF-Main User Defined #2>>[Site] at the <<CF-Main User Defined #4>>[Number].

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### SIGNATURE AND CONSENT

Before making the decision regarding enrollment in this research, you should have:

- Discussed this study with the study doctor or his/her designee;
- Reviewed the information in this form;
- Had the opportunity to ask any questions you may have.

Your signature below means that you have received this information, have asked the questions you currently have about the research, and have received the answers to those questions. You can print a copy of your signed and dated form from the portal to keep for future reference.

| <b>Participant</b> : By signing this consent form, you indicate that you are voluntarily choosing to take part in this research. | | | |
|---|---|---|---|
| Signature of Participant | Date | Time | Printed Name |
| Person Explaining the Research (Principal Investigator or Designee): Your signature below means that you have explained the research to the participant and have answered any questions about the research. | | | |
| Principal Investigator or Designee | Date | Time | Printed Name |

LEAP-CT for evaluation of post-exposure prophylaxis for newly-infected COVID-19 patients 18 February 2022

IRB Approved Template MUST BE APPROVED FOR SITES BEFORE USE AS MODIFIED Jul 07, 2022

#### PARTICIPATION IN A FOLLOW-ON RESEARCH STUDY

We may contact you in the near future to see if you would like to participate in a potential long-term observational study that will be using the data and information already provided by you. During this year-long study, we would ask you to provide daily or weekly updates on your health post-COVID. Please indicate below if you would like to be contacted in the future to be a part of this study.

Yes, you may contact me about participating in this related research study.

| Yes, you may contact me about participating in this related research study. | | | |
|---|---|---|---|
| No, I do not want to be contacted about this related research study. | | | |
| <br>Signature of Participant | Date | Time | Printed Name |